CLINICAL TRIAL: NCT04202289
Title: Evaluation of Nile Tilapia (Oreochromis Niloticus) Skin as an Occlusive Biological Dressing in the Treatment of Burn Wounds: Phase III Randomized Controlled Trial
Brief Title: Use of Nile Tilapia Fish Skin as a Xenograft for Burn Treatment: Phase III Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara (Other)
Responsible Party: Principal Investigator, Edmar Maciel Lima Júnior, MD, Plastic Surgeon, Nucleo De Pesquisa E Desenvolvimento De Medicamentos Da Universidade Federal Do Ceara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nile Tilapia Fish Skin
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Burns
Keywords: Burns; Nile tilapia; Xenograft; Oreochromis niloticus; Biocompatible materials; Wound healing
MeSH Terms: conditions — Burns | interventions — Silver Sulfadiazine

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, monocentric, open-label, controlled phase III clinical study
Masking Description: Patients were blinded to the hypothesized effects of either treatment, but neither the patients nor the consultant were blinded to the treatment administered, due to the necessity of visualizing the treatments in order to conduct them properly (i.e., both types of dressing need to be seen to be applied, evaluated, replaced and removed adequately).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver Sulfadiazine Cream 1% (Active Comparator): In the control group, after cleaning the lesion with tap water and 2% chlorhexidine gluconate, a thin layer of Silver Sulfadiazine Cream 1% was applied and covered with gauze and bandage. The dressing changes occurred every 48 hours. The patients were evaluated every 48 hours for the study parameters.
  Interventions: Drug: Silver Sulfadiazine Cream 1%
- Nile Tilapia Fish Skin (Experimental): In the test group, the treatment was Nile Tilapia Fish Skin, which have a patent registered at the National Institute of Industrial Property (INPI) under number BR 10 2015 021435 9. Nile Tilapia Fish Skin was subjected to a rigorous process of chemical sterilization, glycerolization and irradiation, followed by microbiological tests for bacteria and fungi, before storage in sterile refrigerated packaging. Prior to its use in the patient, the skin was washed thrice in sterile 0.9% saline for 5 minutes, in order to remove glycerol. Regarding application in the study patients, after cleaning the lesion with tap water and 2% chlorhexidine gluconate, Nile Tilapia Fish Skin was applied and covered with gauze and bandage. Throughout the treatment, dressings with Nile Tilapia Fish Skin were only changed if the biomaterial was not properly adhered to the wound bed. The patients were evaluated every 48 hours for the study parameters.
  Interventions: Device: Nile Tilapia Fish Skin

INTERVENTIONS:
Device: Nile Tilapia Fish Skin — In the search of new therapies for burns, the skin of Brazil's most cultivated fish, the Nile tilapia, which was mostly a waste product (although sometimes used as a resistant material for artisanal handicraft), was suggested as a possibility for the development of a low-cost xenograft. Apart from non-infectious microbiota, Nile Tilapia Fish Skin presented histomorphological similarities with human skin in pre-clinical studies. It was shown to have a deep dermis formed by thick collagen fibers organized on parallel/horizontal and transversal/vertical arrangement and composed, in comparison, by larger amounts of type I collagen. Nile Tilapia Fish Skin did not present variations in its microscopic structure and tensile strength after glycerolization, irradiation and posterior rehydration, recovering its natural consistency after glycerol removal.
  Other Names: Tilapia Skin
  Arms: Nile Tilapia Fish Skin
Drug: Silver Sulfadiazine Cream 1% — Topical antibiotic commonly used for the treatment of superficial and deep partial-thickness burns.
  Other Names: Silver Sulfadiazine
  Arms: Silver Sulfadiazine Cream 1%

SUMMARY:
The present study is a Phase III Randomized Clinical Trial aiming to evaluate the efficacy of Nile tilapia (Oreochromis niloticus) skin as an occlusive biological dressing in the treatment of superficial partial-thickness burns in adults.

DETAILED DESCRIPTION:
This is a prospective, randomized, monocentric, open-label, controlled phase III clinical study conducted in Fortaleza, Brazil, from April 2017 to October 2018. The local Institutional Review Board approved the study protocol and informed consent, which was obtained from all participants. The research was conducted in accordance with the 1975 Declaration of Helsinki and its amendments.

The study population consisted of 115, both male and female, participants, who were recruited from a local burn treatment center. Inclusion criteria were: age ≥ 18 and ≤60 years; the presence of dermatological wounds caused by superficial partial-thickness burns (SPTB) affecting up to 15% of Total Body Surface Area (TBSA) and with indication for outpatient treatment; the absence of previous treatment for the current burn and an absence of other significant diseases that could impact the volunteer's participation in the study (coronary artery disease, peripheral vascular disease, cancer, diabetes mellitus, among others). Exclusion criteria included hypersensitivity to materials used in the study or to related compounds; history of severe adverse reactions; drug addiction, including alcohol; use of medications that could have an impact on wound healing (e.g., steroids) and pregnancy, labor or miscarriage in the 12 weeks before the scheduled start of treatment.

In the test group, the treatment was Nile Tilapia Fish Skin, which have a patent registered at the National Institute of Industrial Property (INPI) under number BR 10 2015 021435 9. Nile Tilapia Fish Skin was subjected to a rigorous process of chemical sterilization, glycerolization and irradiation, followed by microbiological tests for bacteria and fungi, before storage in sterile refrigerated packaging. Prior to its use in the patient, the skin was washed in sterile 0.9% saline for 5 minutes, with this process being repeated three times in a row. In the control group, conventional treatment with silver sulfadiazine cream 1% was applied. Randomization was performed using a predefined computer-generated list, with 57 patients being allocated in the test group and 58 patients being allocated in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤60 years.
* Presence of dermatological wounds caused by superficial partial-thickness burns (SPTB) affecting up to 15% of Total Body Surface Area (TBSA).
* Patient with indication for outpatient treatment.

Exclusion Criteria:

* Previous treatment for the current burn.
* Presence of other significant diseases that could impact the volunteer's participation in the study (coronary artery disease, peripheral vascular disease, cancer, diabetes mellitus, among others).
* Hypersensitivity to materials used in the study or to related compounds.
* History of severe adverse reactions; drug addiction, including alcohol.
* Use of medications that could have an impact on wound healing (e.g., steroids).
* Pregnancy, labor or miscarriage in the 12 weeks before the scheduled start of treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Number of days for complete reepithelialization of the burn wound | Day 11
  Number of days until complete reepithelialization of the burn wound, considering application of the first dressing as day zero. Complete reepithelialization was defined as a ≥95% reepithelialization calculated via clinical judgment from the consultant
Number of dressings performed | Day 11
  In the control group, a dressing change was defined as the act of cleaning the wound and reapplying the Silver Sulfadiazine Cream 1%, which was performed every 48 hours. In the test group, a dressing change was defined as the act of replacing the Nile Tilapia Fish Skin which did not adhere properly and/or replacing gauze and bandage that is full of exudate.
Amount of anesthetics used throughout the treatment | Day 11
  In order to audit analgesic intake, apart from the medication prescription (dipyrone and/or tramadol), the patients received a daily record card. They were asked to take the medication only if they felt pain, always respecting instructions in the prescription, and to register the amount of medication taken and the date on the card. Upon returning for medical evaluation, the remaining medication was checked and compared to the daily record card.
Treatment cost per patient | Day 11
  Consumption of materials of the burn treatment center was controlled by the completion of a specific form, an activity performed at the end of each patient visit by the nursing staff. The resources consumed were divided into three categories: a) products used for wound management (either Nile Tilapia Fish Skin or Silver Sulfadiazine Cream 1%); (b) hospital material required for dressing preparation (such as sterile gloves, chlorhexidine, gauze, and bandage); and c) analgesic medication required throughout treatment (dipyrone and/or tramadol). Human resources were not evaluated.

SECONDARY OUTCOMES:
Pain intensity evaluation via Visual Analogue Scale scores | Day 1, 3, 5, 7, 9 and 11
  Patients were informed that the left end of the 10 cm horizontal line (with a "0") represented "no pain" and that the right end (with a "10") represented the "most severe pain imaginable." They were asked to make a mark on the line that represented their current pain intensity, and the Visual Analogue Scale pain intensity level was scored by measurement of the distance from the mark to the "no pain" end of the line.
Pain intensity evaluation via Electronic von Frey | Day 1, 3, 5, 7, 9 and 11
  In the Electronic von Frey, a rigid tip of 0.7 mm in diameter is connected to an electronic system, which displays the test readings in grams (from 0.1 to 1000 g). Initially, 4 different points around the burn were chosen, each one with a distance of around 1 cm from the wound bed. The tip was applied perpendicularly to the skin surface in each of these points, with the application rate controlled entirely by the observer. The participants gave a verbal signal when the pressure was felt to be unpleasant: this measure was taken as the Mechanical Pain Threshold of that point. Subsequently, the process was repeated in a similar region of the contralateral healthy side of the body. The mean of the measures of the 4 points in each area was taken as the mean Mechanical Pain Threshold of that area. Finally, the difference between the nociception threshold of healthy skin and of the edge of the burn, expressed in grams, was determined.
Burns Specific Pain Anxiety Scale (BSPAS) scores | Day 5 and 11
  The Brazilian version of the 9-item Burns Specific Pain Anxiety Scale (BSPAS) was employed. Each item in the BSPAS is scored on a 10 cm visual analogue line with two reference points given values of 0 and 10. The patient is asked how much the assertions relate to their current pain situation, with 0 corresponding to ''not at all'' and 10 corresponding to ''the worst imaginable way''. The total score is calculated by adding up the scores for all items, with a maximum of 90 points.
Burn improvement on the day of dressing removal evaluation | Day 11
  Assessed via the Clinical Global Impression Scale-Improvement (CGI-I). The CGI-I is evaluated by the physician responsible and answers the following question: "Compared to the patient's condition at admission to the project, this patient's condition is: 1 - very much improved since the initiation of treatment; 2 - much improved; 3 - minimally improved; 4 - no change from baseline; 5 - minimally worse; 6 - much worse; 7 - very much worse since the initiation of treatment".

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisabete A de Moraes, MD, PhD, Study Director — Drug Research and Development Center (NPDM)
Locations (2):
- Brazil (2):
  - Burn Treatment Center, Dr. José Frota Institute, Fortaleza, Ceará
  - Drug Research and Development Center (NPDM), Federal University of Ceará (UFC), Fortaleza, Ceará

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lima-Junior EM, de Moraes Filho MO, Costa BA, Fechine FV, de Moraes MEA, Silva-Junior FR, Soares MFADN, Rocha MBS, Leontsinis CMP. Innovative treatment using tilapia skin as a xenograft for partial thickness burns after a gunpowder explosion. J Surg Case Rep. 2019 Jun 14;2019(6):rjz181. doi: 10.1093/jscr/rjz181. eCollection 2019 Jun. PMID 31214319
- [Background] Costa BA, Lima Junior EM, de Moraes Filho MO, Fechine FV, de Moraes MEA, Silva Junior FR, do Nascimento Soares MFA, Rocha MBS. Use of Tilapia Skin as a Xenograft for Pediatric Burn Treatment: A Case Report. J Burn Care Res. 2019 Aug 14;40(5):714-717. doi: 10.1093/jbcr/irz085. PMID 31112268
- [Background] Lima Junior EM, Moraes Filho MO, Forte AJ, Costa BA, Fechine FV, Alves APNN, Moraes MEA, Rocha MBS, Silva Junior FR, Soares MFADN, Bezerra AN, Martins CB, Mathor MB. Pediatric Burn Treatment Using Tilapia Skin as a Xenograft for Superficial Partial-Thickness Wounds: A Pilot Study. J Burn Care Res. 2020 Feb 19;41(2):241-247. doi: 10.1093/jbcr/irz149. PMID 31504615
- [Background] Alves APNN, Lima Junior EM, Piccolo NS, de Miranda MJB, Lima Verde MEQ, Ferreira Junior AEC, de Barros Silva PG, Feitosa VP, de Bandeira TJPG, Mathor MB, de Moraes MO. Study of tensiometric properties, microbiological and collagen content in nile tilapia skin submitted to different sterilization methods. Cell Tissue Bank. 2018 Sep;19(3):373-382. doi: 10.1007/s10561-017-9681-y. Epub 2018 Jan 29. PMID 29380095
- See also: Register on ClinicalTrials.gov of the Phase II Randomized Controlled Trial evaluating the use of Tilapia Skin in the treatment of burn wounds. — https://clinicaltrials.gov/ct2/show/NCT03592498